CLINICAL TRIAL: NCT04150185
Title: Prospective Comprehensive Assessment of Quality of Life and Psychology After Donor Hepatectomy
Brief Title: Quality of Life and Psychology of Donors After Hepatectomy
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Piyush Kumar Sinha, Assistant Professor Liver Transplant Surgery, Institute of Liver and Biliary Sciences, India
Other Study IDs: f25/5/15/AC/ILBS/2011/213
Record Dates: First submitted 2019-10-28; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- live liver donors: Live liver donors undergoing donor hepatectomy
  Interventions: Procedure: Donor hepatectomy

INTERVENTIONS:
Procedure: Donor hepatectomy

SUMMARY:
Liver donation by a living donor is major surgery and has a profound effect on health-related quality of life and psychology. This study aims at evaluating those aspects of a donor for a period of five years after surgery.

DETAILED DESCRIPTION:
Live donor liver transplantation (LDLT) has established itself as a treatment for end-stage liver disease but donor safety remains a major issue. It is the responsibility of the transplant team to restore donor's health, not only physical, but also mental, social and environmental. There is scarcity of long term longitudinal data on donor quality of life. Most of the studies are cross sectional which describe the quality of life at certain time point and do not take into account of changes that might occur over a period. It is more relevant in this scenario, as two persons from a family undergo surgery at the same time, which has a profound effect on family dynamics, and restoration towards normalcy goes hand in hand with adaptation to a new lifestyle. Another shortcoming of available literature is lack of uniform instruments which comprehensively measure the quality of life of live liver donors (LLDs). Standardized health related quality of life (HRQOL) instruments such as Short Form 36(SF 36) or World Health Organization quality of life Brief (WHOQOL-BREF) are not designed for LLDs. Moreover, there are several symptoms which might interfere with daily activities such as incision site problems , dyspepsia to name a few, but are not distressing enough to be reflected on quality of life scores .The aim of current study was to observe the attitude of donors pre transplant, quality of life over a period, satisfaction with the donation process, their assessment of the health care team, satisfaction with the consent process, and change in pattern of symptoms and cosmesis after surgery.

ELIGIBILITY:
Inclusion Criteriteria:

- All patients undergoing donor hepatectomy from March 2012 to August 2013

Exclusion Criteria:

- Refusal to participate in study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All donors undergoing donor hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Health Related quality of life: WHOQOL Bref Hindi | Predonation and at 1week,1 month, 3 months, 1 year,2 year,3 year, 5 year
  Health related quality of life measured using World Health Organization Quality of Life Brief in hindi language. There are 4 domains namely physical, psychological, social and environmental.The scores in each domain vary from 0 to 100 with higher score means better.

SECONDARY OUTCOMES:
cosmetic score | Predonation and at 1week,1 month, 3 months, 1 year,2 year,3 year, 5 year
  The body image and cosmesis questionnaire consists of eight questions combined to form two scales: a body image scale and a cosmesis scale. Five questions regarding body image assess patient's perception of their own body and their satisfaction with that perception, while also evaluating patient's attitude toward their bodily appearance. The body image scale ranges from 5 (lowest body image score) to 20 (highest body image score). Three questions regarding the cosmetic result after the operation assess the degree of satisfaction with respect to the physical appearance of the incisional scar. The combined scores of these three questions resulted in the cosmesis scale ranging from 3 (lowest satisfaction) to 24 (highest satisfaction)
body weight | Predonation and at 1week,1 month, 3 months, 1 year,2 year,3 year, 5 year
  weight of donors
financial status | before donation and after 2 years
  annual income
donor symptoms questions | Predonation and at 3 months, 1 year,2 year,3 year, 5 year
  These questions were based on the long term effect of cholecystectomy, incision site problems and abdominal surgery in general. The questions included gastro esophageal reflux disease (GERD)/Heartburn, nausea/vomiting, incision site discomfort and alteration in bowel habit. The number of donors reporting these symptoms were assessed to calculate the incidence at predefined time points.

CONTACTS AND LOCATIONS:
Overall Officials: Piyush K Sinha, MS, MCh, Principal Investigator — Assistant Professor, liver transplant surgery

IPD SHARING:
Plan to Share IPD: No